CLINICAL TRIAL: NCT00037505
Title: Major Depression and Inflammatory Risk Markers for Coronary Heart Disease
Status: Completed | Type: Observational
Sponsor: National Center for Research Resources (NCRR) (NIH)
Collaborators: American Heart Association (Other)
Other Study IDs: NCRR-M01RR00036-0849
Record Dates: First submitted 2002-05-17; First posted 2002-05-20 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2003-12

CONDITIONS: Depression
MeSH Terms: conditions — Depression

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Other

SUMMARY:
The overall purpose of this research is to examine whether depression influences immune system function. Studies indicate that individuals who are depressed experience coronary heart disease at a higher rate than expected. This study's goal is to begin identifying mechanisms that might be responsible for this process. This research also examines whether behavioral processes (e.g. smoking) or hormonal processes (e.g. adrenaline release) are responsible for immune system differences between depressed and nondepressed people

DETAILED DESCRIPTION:
To qualify for participation, subjects are to be between the ages of 18-55, medically healthy and free of all medication three months prior to enrollment. Half of them will be clinically depressed; the remaining one half will be healthy controls without a history of psychiatric illness. All subjects who qualify for the study will attend two laboratory sessions. During the first visit, participants will undergo a structured psychological interview, complete questionnaires about their mood, personality, and behavior, and have blood drawn to assess their immune system function. During the second visit, participants will complete additional questionnaires about their mood, personality, and behavior. The subjects will also participate in a mock job interview to look at their body's response to stress. Before and after the interview, the subjects will have blood drawn and be asked to collect saliva samples to assess their immune system function. In addition to the two laboratory visits, participants will be asked to collect additional information while going about their normal activities. In order to accomplish this, they will be given a small hand held portable computer. Four times each day for four days, the computer will signal them to collect a saliva sample. This will be used later to measure hormone levels. This study will explore changes in the immune system and metabolic system that might predispose depressed individuals to develop heart disease

ELIGIBILITY:
For eligibility, potential subjects will be 18-55 years of age, free of all medication during the past three months, and have no history of chronic illness involving the cardiovascular, endocrine, immune systems

Ages: 15 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult

CONTACTS AND LOCATIONS:
Locations (1):
- Washington University, St Louis, Missouri, United States